CLINICAL TRIAL: NCT04353141
Title: A Prospective International Lung UltraSound Analysis (ILUSA) Study in Tertiary Maternity Wards During the SARS-CoV-2 Pandemic
Brief Title: International Lung UltraSound Analysis (ILUSA) Study
Acronym: ILUSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Dirk Timmerman, PhD, KU Leuven
Other Study IDs: COVID-19: ILUSA (S63988)
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: COVID; Pregnancy Complications, Infectious; Pregnancy Related; Pregnancy, High Risk; Pregnancy Disease; Pneumonia; Pneumonia, Viral; Diagnoses Disease
Keywords: COVID-19; Pregnancy; Diagnosis; Lung ultrasound; Pneumonia; Oxygen support
MeSH Terms: conditions — Pregnancy Complications, Infectious; Pneumonia; Pneumonia, Viral; COVID-19; Disease | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnant patients with confirmed COVID-19 infection
  Interventions: Diagnostic Test: standardized Lung Ultrasound (LUS) examination
- Pregnant patients symptomatic for COVID-19: Symptomatic patients suspicious for COVID-19 infection (swab is taken on admission)
  Interventions: Diagnostic Test: standardized Lung Ultrasound (LUS) examination
- Pregnant patients asymptomatic for COVID19: Patients asymptomatic for COVID19 with other feto-maternal diseases or who come for delivery or caesarean section
  Interventions: Diagnostic Test: standardized Lung Ultrasound (LUS) examination

INTERVENTIONS:
Diagnostic Test: standardized Lung Ultrasound (LUS) examination — 14 areas (three posterior, two lateral and two anterior) will be assigned a COVID-LUS score: Score 0 (Normal pattern), Score 1 (Pattern of mild disease), Score 2 (Pattern of moderate disease), Score 3 (Pattern of severe disease). Classification of LUS result: LUS NEGATIVE: Group A = Score 0 in all 14 areas OR score =1 in areas of one site (right or left). It means that score 1 is pathological only when present bilaterally; LUS POSITIVE: both group B and C have to be considered positive: Group B (MILD DISEASE) = Score 1 in at least two areas localized bilaterally and no areas with score >1; Group C (MODERATE/SEVERE DISEASE)= Score >2 in at least two areas localized bilaterally

SUMMARY:
Currently there is a great need for an accurately and rapid assessment of patients suspected for Covid-19. Like CT, Lung Ultrasound (LUS) examination can potentially help with the initial triage of patients but also help track the evolution of the disease. LUS can be used in every setting, including settings with limited infrastructure, allowing the reduction of disparities in trials participation. LUS is also a practical approach that can be used by obstetricians/gynecologists, who are the primary care givers in the labour and delivery room.

The International Lung UltraSound Analysis (ILUSA) Study is an international multicenter prospective explorative observational study to assess the predictive value of LUS in Covid-19 suspected and diagnosed pregnant patients.

DETAILED DESCRIPTION:
During the current COVID-19 outbreak, all patient groups have been affected, also the most fragile such as the pregnant women. Although experts provided general suggestions on the best management of pregnant women with suspected or confirmed COVID-19, these considerations are mainly based on retrospective studies or case series. No prospective study is currently available about management of confirmed or suspected patients during pregnancy. Moreover, only limited outcome data is available on the management of asymptomatic SARS-CoV-2 positive pregnant patients, many of whom subsequently develop disease symptoms.

The current gold standard for the etiological diagnosis of COVID-19 infection is analysis of respiratory tract specimens by (real-time) reverse transcription polymerase chain reaction (RT-PCR). However, this test has a high false-negative rate, due to both nasopharyngeal swab sampling error, which often requires repeat sampling, and changing viral burden. Currently, high-resolution computed tomography (CT) is the main tool for primary diagnosis and evaluation of disease severity in patients affected by COVID-19 infection. Chest CT scan also demonstrated a specificity even superior to the nasal/pharyngeal swab for diagnosis. Yet, radiation exposure should ideally be avoided at all times in pregnancy. A radiation-free point-of-care diagnostic tool, such as lung ultrasound (LUS) examination, would be particularly useful for assessing the lungs of pregnant women. Indeed, LUS examination has recently been suggested by the Chinese Critical Care Ultrasound Study Group and the Italian Academy of Thoracic Ultrasound as an accurate tool to detect lung involvement during COVID-19.

In pregnant patients, LUS could be a valid alternative imaging tool to thoracic CT to guarantee appropriate care for these patients. Symptomatic patients with a low risk of developing serious disease may be possibly reassured, and could leave the hospital soon after delivery. On the other hand LUS could possibly indicate patients at higher risk for future need of oxygen or ventilation support, and who might need more careful monitoring and longer hospitalization. In view of the wide availability in delivery suites, the low cost and easy bedside application LUS could also be readily repeated during patient follow up as needed. LUS has been traditionally employed by non-radiologists as an adjunctive clinical instrument. Obstetricians represent a category of clinicians who use ultrasound in their daily routine practice. From a technical point of view, examination of the lungs at the time of obstetric ultrasound evaluation could be feasible for obstetricians and gynaecologists.

Currently there is a great need for an accurately and rapid assessment of patients suspected for Covid-19. Like CT, LUS can potentially help with the initial triage of patients but also help track the evolution of the disease. LUS can be used in every setting, including settings with limited infrastructure, allowing the reduction of disparities in trials participation. LUS is also a practical approach that can be used by obstetricians/gynecologists, who are the primary care givers in the labour and delivery room.

The International Lung UltraSound Analysis (ILUSA) Study is an international multicenter prospective explorative observational study to assess the predictive value of LUS in Covid-19 suspected and diagnosed pregnant patients.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this Trial must meet all of the following criteria:

Voluntary written informed consent of the participant or their legally authorized representative obtained prior to any screening procedures

Pregnant patients admitted to the Hospital during the COVID-19 pandemic:

1. Patients with confirmed COVID-19 infection (see below)
2. Symptomatic patients suspicious for COVID-19 infection (swab is taken on admission)
3. Patients asymptomatic for COVID19 with other feto-maternal diseases or who come for delivery or caesarean section

All participants that are considered for Trial participation, per the above criteria will be documented on the Screening Log, including Screen Failures.

Definition of suspected case (WHO guideline, ISUOG)

1. A patient with acute respiratory illness (fever and at least one sign/symptom of respiratory disease (e.g. cough, shortness of breath)) AND with no other etiology that fully explains the clinical presentation AND a history of travel to or residence in a country/area or territory reporting local transmission of COVID-19 infection during the 14 days prior to symptom onset; OR
2. A patient with any acute respiratory illness AND who has been in contact with a confirmed or probable case of COVID-19 infection in the 14 days prior to onset of symptoms; OR
3. A patient with severe acute respiratory infection (fever and at least one sign/symptom of respiratory disease (e.g. cough, shortness breath)) AND who requires hospitalization AND who has no other etiology that fully explains the clinical presentation.

Exclusion Criteria:

Participants eligible for this Trial must not meet any of the following criteria:

* Maternal lung pre-existing disease
* Maternal cardiac problems
* Severely ill patients in unstable condition requiring immediate life-saving procedures

Participants who meet one or more of the above exclusion criteria must not proceed to be enrolled in the Trial and will be identified on the Screening Log as Screen Failure.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive pregnant patients who are admitted to the hospital for delivery, cesarean section or admission for at least one night.
Sampling Method: Probability Sample
Enrollment: 1850 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of LUS to predict poor outcome | outcome one week after enrollment into the study
  The primary endpoint is diagnostic performance in terms of the area under the receiver operating characteristic curve (AUC, also known as the c-statistic) and sensitivity and specificity with regard to the prediction of poor outcome.
  Outcome at one week from admission: good outcome includes discharge or inpatient breathing in free air; poor outcome includes patient with oxygen support, patients with CPAP/ high oxygen flow cannula, or patient with endotracheal intubation during the week.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Timmerman, PhD, Study Chair — KU Leuven, Leuven BE; Antonia Testa, PhD, Study Chair — Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Rome IT; Jan Deprest, PhD, Study Chair — KU Leuven; Francesca Moro, MD, Study Chair — Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Rome IT; Tom Bourne, PhD, Study Chair — Queen Charlotte's & Chelsea Hospital, Imperial College London, London, UK; Giovanni Scambia, PhD, Study Chair — Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Rome IT; Antonio Lanzone, PhD, Study Chair — Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Rome IT
Locations (7):
- University Hospitals Leuven, Leuven, Belgium
- Italy (5):
  - University of Brescia, Brescia
  - University of Foggia, Foggia
  - University of Milan, Milan
  - University of Parma, Parma
  - Fondazione Policlinico Universitario A. Gemelli, Roma
- Queen Charlotte's & Chelsea Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen H, Guo J, Wang C, Luo F, Yu X, Zhang W, Li J, Zhao D, Xu D, Gong Q, Liao J, Yang H, Hou W, Zhang Y. Clinical characteristics and intrauterine vertical transmission potential of COVID-19 infection in nine pregnant women: a retrospective review of medical records. Lancet. 2020 Mar 7;395(10226):809-815. doi: 10.1016/S0140-6736(20)30360-3. Epub 2020 Feb 12. PMID 32151335
- [Background] Liu D, Li L, Wu X, Zheng D, Wang J, Yang L, Zheng C. Pregnancy and Perinatal Outcomes of Women With Coronavirus Disease (COVID-19) Pneumonia: A Preliminary Analysis. AJR Am J Roentgenol. 2020 Jul;215(1):127-132. doi: 10.2214/AJR.20.23072. Epub 2020 Mar 18. PMID 32186894
- [Background] Schwartz DA. An Analysis of 38 Pregnant Women With COVID-19, Their Newborn Infants, and Maternal-Fetal Transmission of SARS-CoV-2: Maternal Coronavirus Infections and Pregnancy Outcomes. Arch Pathol Lab Med. 2020 Jul 1;144(7):799-805. doi: 10.5858/arpa.2020-0901-SA. PMID 32180426
- [Background] Mullins E, Evans D, Viner RM, O'Brien P, Morris E. Coronavirus in pregnancy and delivery: rapid review. Ultrasound Obstet Gynecol. 2020 May;55(5):586-592. doi: 10.1002/uog.22014. PMID 32180292
- [Background] Liu Y, Chen H, Tang K, Guo Y. Withdrawn: Clinical manifestations and outcome of SARS-CoV-2 infection during pregnancy. J Infect. 2020 Mar 5:S0163-4453(20)30109-2. doi: 10.1016/j.jinf.2020.02.028. Online ahead of print. PMID 32145216
- [Background] Poon LC, Yang H, Lee JCS, Copel JA, Leung TY, Zhang Y, Chen D, Prefumo F. ISUOG Interim Guidance on 2019 novel coronavirus infection during pregnancy and puerperium: information for healthcare professionals. Ultrasound Obstet Gynecol. 2020 May;55(5):700-708. doi: 10.1002/uog.22013. Epub 2020 Mar 20. No abstract available. PMID 32160345
- [Background] Rasmussen SA, Smulian JC, Lednicky JA, Wen TS, Jamieson DJ. Coronavirus Disease 2019 (COVID-19) and pregnancy: what obstetricians need to know. Am J Obstet Gynecol. 2020 May;222(5):415-426. doi: 10.1016/j.ajog.2020.02.017. Epub 2020 Feb 24. PMID 32105680
- [Background] Liang H, Acharya G. Novel corona virus disease (COVID-19) in pregnancy: What clinical recommendations to follow? Acta Obstet Gynecol Scand. 2020 Apr;99(4):439-442. doi: 10.1111/aogs.13836. Epub 2020 Mar 5. No abstract available. PMID 32141062
- [Background] Hao W, Li M. Clinical diagnostic value of CT imaging in COVID-19 with multiple negative RT-PCR testing. Travel Med Infect Dis. 2020 Mar-Apr;34:101627. doi: 10.1016/j.tmaid.2020.101627. Epub 2020 Mar 13. No abstract available. PMID 32179123
- [Background] Pan Y, Guan H, Zhou S, Wang Y, Li Q, Zhu T, Hu Q, Xia L. Initial CT findings and temporal changes in patients with the novel coronavirus pneumonia (2019-nCoV): a study of 63 patients in Wuhan, China. Eur Radiol. 2020 Jun;30(6):3306-3309. doi: 10.1007/s00330-020-06731-x. Epub 2020 Feb 13. PMID 32055945
- [Background] Bernheim A, Mei X, Huang M, Yang Y, Fayad ZA, Zhang N, Diao K, Lin B, Zhu X, Li K, Li S, Shan H, Jacobi A, Chung M. Chest CT Findings in Coronavirus Disease-19 (COVID-19): Relationship to Duration of Infection. Radiology. 2020 Jun;295(3):200463. doi: 10.1148/radiol.2020200463. Epub 2020 Feb 20. PMID 32077789
- [Background] Zu ZY, Jiang MD, Xu PP, Chen W, Ni QQ, Lu GM, Zhang LJ. Coronavirus Disease 2019 (COVID-19): A Perspective from China. Radiology. 2020 Aug;296(2):E15-E25. doi: 10.1148/radiol.2020200490. Epub 2020 Feb 21. PMID 32083985
- [Background] Fang Y, Zhang H, Xie J, Lin M, Ying L, Pang P, Ji W. Sensitivity of Chest CT for COVID-19: Comparison to RT-PCR. Radiology. 2020 Aug;296(2):E115-E117. doi: 10.1148/radiol.2020200432. Epub 2020 Feb 19. No abstract available. PMID 32073353
- [Background] Peng QY, Wang XT, Zhang LN; Chinese Critical Care Ultrasound Study Group (CCUSG). Findings of lung ultrasonography of novel corona virus pneumonia during the 2019-2020 epidemic. Intensive Care Med. 2020 May;46(5):849-850. doi: 10.1007/s00134-020-05996-6. Epub 2020 Mar 12. No abstract available. PMID 32166346
- [Background] Soldati G, Smargiassi A, Inchingolo R, Buonsenso D, Perrone T, Briganti DF, Perlini S, Torri E, Mariani A, Mossolani EE, Tursi F, Mento F, Demi L. Is There a Role for Lung Ultrasound During the COVID-19 Pandemic? J Ultrasound Med. 2020 Jul;39(7):1459-1462. doi: 10.1002/jum.15284. Epub 2020 Apr 7. No abstract available. PMID 32198775
- [Background] Buonsenso D, Pata D, Chiaretti A. COVID-19 outbreak: less stethoscope, more ultrasound. Lancet Respir Med. 2020 May;8(5):e27. doi: 10.1016/S2213-2600(20)30120-X. Epub 2020 Mar 20. No abstract available. PMID 32203708
- [Background] Soldati G, Smargiassi A, Inchingolo R, Buonsenso D, Perrone T, Briganti DF, Perlini S, Torri E, Mariani A, Mossolani EE, Tursi F, Mento F, Demi L. Proposal for International Standardization of the Use of Lung Ultrasound for Patients With COVID-19: A Simple, Quantitative, Reproducible Method. J Ultrasound Med. 2020 Jul;39(7):1413-1419. doi: 10.1002/jum.15285. Epub 2020 Apr 13. PMID 32227492
- [Background] Moro F, Buonsenso D, Moruzzi MC, Inchingolo R, Smargiassi A, Demi L, Larici AR, Scambia G, Lanzone A, Testa AC. How to perform lung ultrasound in pregnant women with suspected COVID-19. Ultrasound Obstet Gynecol. 2020 May;55(5):593-598. doi: 10.1002/uog.22028. PMID 32207208